CLINICAL TRIAL: NCT04568746
Title: Impact of the Implementation of a qSOFA Score on the Care of Adult Patients Referred to the Emergency Department for Suspected Infection
Brief Title: Implementation of a qSOFA Score in the Emergency Department
Acronym: qSOFA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: P/2019/452
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Sepsis
Keywords: screening; qSOFA; sepsis; Emergency care unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with qSOFA ≥ 2 (Other): adult patients with a qSOFA score ≥ 2 at the screening in the emergency department, will be referred to the emergency vital room
  Interventions: Procedure: emergency vital room
- patients with qSOFA <2 (Other): adult patients with a qSOFA score < 2 at the screening in the emergency department, will be referred to the box
  Interventions: Procedure: box

INTERVENTIONS:
Procedure: emergency vital room — At the arrival of the patient, the qSOFA will be carried out to guide the orientation. Patient with score ≥ 2 will be supported in emergency vital room
  Arms: patients with qSOFA ≥ 2
Procedure: box — patient with score < 2 will be supported in box
  Arms: patients with qSOFA <2

SUMMARY:
The Quick-SOFA score (qSOFA), identifies septic patients with a mortality risk higher than 10%. In our study all adult patients coming to the emergency for suspected infection are screened according to the qSOFA score on arrival. If qSOFA ≥ 2, the patient should be referred to emergency vital room, if the score <2, the patient will be in the box. The objectives are : 1) to evaluate the mortality at 28 days with the orientation, 2) to compare support time of medical contact and initiation of antibiotics according to the orientation in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* body temperature below 36 °C or above 38 °C
* require hospitalization

Exclusion Criteria:

* hospital transfer,
* patients with pre hospital care
* language barrier,
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
mortality rate | 28 days
  compare mortality rate with orientation in emergency

SECONDARY OUTCOMES:
support time to medical contact | 1 day
  compare support time with orientation of patients according to the orientation of the patient in the emergency department
support time to initiation of antibiotics | 1 day
  compare support time with initiation antibiotics of patients according to the orientation of the patient in the emergency department

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Besancon, Besançon, France